CLINICAL TRIAL: NCT00390754
Title: Utility of Home Pregnancy Testing in Medicaid Women at Risk for Unintended Pregnancy
Brief Title: Usefulness of Home Pregnancy Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Michigan Department of Community Health (Other)
Responsible Party: Mary Nettleman, MD, MS, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 95530-00
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Fertility
Keywords: pregnancy; unintended; menses
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregnancy Test Group (Experimental): Group got free home pregnancy test kits
  Interventions: Behavioral: Education for pregnancy planning
- 2 (No Intervention): Group did not receive free home pregnancy test kits

INTERVENTIONS:
Behavioral: Education for pregnancy planning — Provision of free home pregnancy tests to women at risk for unintended pregnancy
  Other Names: Home pregnancy testing
  Arms: Pregnancy Test Group

SUMMARY:
The objective of this study is to determine whether women in a Medicaid population at risk for unintended pregnancy will keep a home pregnancy test on hand and (if necessary) use it appropriately.

DETAILED DESCRIPTION:
Once pregnancy is recognized, most women seek prompt prenatal care and try to stop risk behaviors. Unfortunately, women with unintended pregnancies do not recognize their pregnancies promptly, and inadvertently continue risk behaviors into the vulnerable early pregnancy weeks. Home pregnancy testing is a rapid and inexpensive means of pregnancy diagnosis. The objective of this study is to determine whether women in a Medicaid population at risk for unintended pregnancy will keep a home pregnancy test on hand and (if necessary) use it appropriately

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 34 year old female,
* sexually active,
* not pregnant,
* not desiring pregnancy,
* not surgically sterile,
* intercourse at least once in the past 6 months without using effective contraception (hormonal or barrier or male vasectomy)
* receiving Medicaid OR child on Medicaid OR Medicaid paid for prev. preg
* understands written/spoken English enough to give informed consent and respond to survey

Exclusion Criteria:

* fails to meet inclusion criteria

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of episodes of use of home pregnancy test kits | 6 month followup

SECONDARY OUTCOMES:
Knowledge about use of home pregnancy test kits | 6 months
Episodes of pregnancy suspicion | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary D. Nettleman, MD, MS, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

REFERENCES:
- [Derived] Nettleman MD, Brewer JR, Ayoola AB. Self-testing for pregnancy among women at risk: a randomized controlled trial. Am J Prev Med. 2009 Feb;36(2):150-3. doi: 10.1016/j.amepre.2008.09.023. Epub 2008 Dec 5. PMID 19062238